CLINICAL TRIAL: NCT02628496
Title: Confocal Laser Microlaryngoscopy (CLMx): A Novel Tool for Noninvasive Evaluation of Laryngeal Lesions
Brief Title: Confocal Laser Microlaryngoscopy (CLMx)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lost funding/staff
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201503127
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Laryngeal Dysplasia; Laryngeal Neoplasm
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Fluorescein; Fluoresceins; Biopsy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: CLM (Experimental): * On the day of surgery, participants will have placement of laser-safe endotracheal tube and a rigid laryngoscope will be introduced into the oral cavity to gain access to the laryngeal introitus and then placed into suspension (standard of care)
  * Fluorescein dye will be administered intravenously
  * Confocal laser probe will be introduced through the rigid laryngoscope and touched first on the lesion of concern and put into scanning mode in order to obtain photos and video footage of the lesions. The probe will then be placed on normal appearing vocal fold tissue to obtain a control sample.
  * The remainder of the procedure is standard excisional biopsy and KTP laser photoablation
  Interventions: Drug: Fluorescein injection, USP 10%; Device: Confocal laser microlaryngoscopy; Procedure: Biopsy (standard of care); Procedure: KTP laser photoablation (standard of care)

INTERVENTIONS:
Drug: Fluorescein injection, USP 10% — -2.5 ml intravenous 10 minutes before procedure
  Other Names: AK-FLUOR
Device: Confocal laser microlaryngoscopy
  Other Names: CLM; CLMx
Procedure: Biopsy (standard of care)
Procedure: KTP laser photoablation (standard of care)

SUMMARY:
The purpose of this study is to evaluate the accuracy and efficacy of using confocal laser microlaryngoscopy (CLM) as a tool to perform non-invasive, in vivo, real time pathologic assessment of laryngeal lesions.

In order to achieve this purpose, this study will prospectively enroll patients with clinical evident laryngeal pathology concerning for cancer or dysplasia, who are scheduled to undergo a formal intraoperative biopsy of their lesion. While in the operating room, prior to performing a formal biopsy, CLM will be used to evaluate the area of pathology, surrounding tissue, and contralateral normal tissue. Then the biopsy will be performed, as per standard protocol, and the diagnostic results from CLM and the formal biopsy will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be adults 18 years of age or older who present to clinic with a history of hoarseness and voice changes and are noted to have changes to their vocal folds that are concerning for the possibility of dysplasia or early stage malignancy.
* Patient will have vocal fold leukoplakia or other abnormal epithelial changes.
* Patient (or legally authorized representative) must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patient must not have a history of radiation to the neck.
* Patient must not have a documented reaction to fluorescein
* Patient must not have a previous history of laryngeal cancer.
* Patient must not have a history of allergy or bronchial asthma.
* Patient must not be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the CLM as measured by the proportion of dysplasia cases that are correctly identified by the probe | Day of surgery (Day 1)
Specificity of the CLM as measured by the proportion of patients with neoplasm cases correctly identified by the probe | Day of surgery (Day 1)
Accuracy of the CLM as measured by the proportion of cases correctly classified by the probe | Day of surgery (Day 1)
  -If the prevalence of the disease in the population is known, the accuracy of the test can be calculated bases on prevalence sensitivity, specificity using the formula: Sensitivity*Prevalence + Specificity*(1-Prevalence)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bradley, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu